CLINICAL TRIAL: NCT04248478
Title: The Relationship Between Eating Behaviours and Health Status of Female Patients With Fibromyalgia
Brief Title: Eating Behaviours in Female Patients With Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Collaborators: Mehmet Akif Ersoy Canakkale State Hospital (Other Government)
Responsible Party: Principal Investigator, Alper Mengi, Medical Doctor, Physiatrist, Gaziosmanpasa Research and Education Hospital
Other Study IDs: KAEK-27/2020-2000006994
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Eating Behavior; Fibromyalgia; Health Status
Keywords: Chronic Pain; Eating Habits
MeSH Terms: conditions — Feeding Behavior; Fibromyalgia; Chronic Pain | interventions — Health Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromiyalgia Patients: Patients diagnosed with fibromyalgia according to 2013 American College of Rheumatology criteria are planned to be included in this arm.
  Interventions: Other: Eating Behaviours; Other: Health Status
- Healthy Volunteers: Healthy volunteers are planned to be included in this arm.
  Interventions: Other: Eating Behaviours

INTERVENTIONS:
Other: Eating Behaviours — Patients' eating behaviour will be questioned with Three Factor Eating Questionnaire. The 18-item Three-Factor Eating Questionnaire is a scale that measures three domains of eating behavior: cognitive restraint , uncontrolled eating and emotional eating.
Other: Health Status — The effect of fibromyalgia on the daily life of the patients will be questioned with Fibromyalgia Impact Questionnaire (FIQ). The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week.
  Groups: Fibromiyalgia Patients

SUMMARY:
The Relationship Between Eating Behaviours and Health Status of Female Patients with Fibromyalgia

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the nutritional behaviours of female patients with fibromyalgia according to the healthy population and the relationship of these behaviours with the current health status of the patient.

In the investigatgor's clinical practice, eating-related problems (increased or decreased appetite, uncontrolled eating, etc.) are observed in fibromyalgia patients. In this study, it will be investigated whether this situation is different from healthy population and whether it is related with the healt status.

Patients diagnosed with fibromyalgia according to 2013 American College of Rheumatology criteria and healthy volunteers are planned to be included in the study.

Demographic data (sex, age, level of education, job, socio-economic situation) will be questioned and their body mass indexes (BMI) will be calculated from all participitants All participants' eating behaviour will be questioned with Three Factor Eating Questionnaire.

In fibromyalgia patients, effect of fibromyalgia on the daily life of the patients will be questioned with Fibromyalgia Impact Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between the ages of 18-40
* Patients diagnosing fibromyalgia for the first time according by 2013 American College of Rheumatology (ACR) criteria

Exclusion Criteria:

* History of eating disorders such as anorexia nervosa, bulimia nevroza
* History of hypothyroidism or hyperthyroidism
* Pregnant or breast feeding
* History of central or peripheral nervous system disorders
* History of infectious, chronic inflammatory disease, malignant tumors
* Subjects with active psychiatric illness or who use psychiatric medication
* Uncooperative subject
* History of cardiac pathology such as heart failure, coronary artery disease
* History of diabetes, chronic renal insufficiency, chronic liver failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients diagnosed with fibromyalgia and healthy volunteers are planned to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
eating behaviour | 7 days
  Participants' eating behaviour will be questioned with Three Factor Eating Questionnaire (TFEQ). The TFEQ contains 51 items (questions) and measures three dimensions of human eating behavior 'cognitive restraint of eating' (Factor I - 21 items) 'disinhibition' (Factor II - 16 items) 'hunger' (Factor III - 14 items). Each item scores either 0 or 1 point. The minimum score for factors I-II-III is therefore 0-0-0, the possible maximum score 21-16-14.

SECONDARY OUTCOMES:
activities of daily living | 7 days
  The effect of fibromyalgia on the daily life of the patients will be questioned with Fibromyalgia Impact Questionnaire (FIQ). The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures 10 items (physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being) over the past week. The maximum possible score of each subtitle is 10. Thus, the total maximum score is 100, a lower score indicates better quality of life.
body mass index | 1 day
  The participants' weights and heights will be measured and the body mass index will be calculated from the measured values.
sex | 1 day
  It will be registered as male or female.
age | 1 day
  The age of the participant will be recorded.
level of education | 1 day
  The education status will be recorded as not literate, primary school, secondary school, high school or university.
job | 1 day
  The job will be recorded as unemployed, housewife, office worker or heavy duty worker.
socio-economic situation | 1 day
  Socio-economic situation will be recorded as income less than expense, income equal to expense or income lower than expense.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Mengi, M.D., Principal Investigator — Canakkale State Hospital
Locations (1):
- Alper Mengi, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No